CLINICAL TRIAL: NCT03893682
Title: A Phase Ia/b Trial to Evaluate the Safety and Tolerability of CG-806 in Patients With CLL/SLL or Non-Hodgkin's Lymphomas
Brief Title: A Study of CG-806 in Patients With Relapsed or Refractory CLL/SLL or Non-Hodgkin's Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in corporate strategy
Sponsor: Aptose Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APTO-CG-806-01
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Oral; DLBCL; PMBCL; BCLU; GZL; MCL; FL; MZL; WM; LPL; CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): CG-806 will be given orally in ascending doses in patients with relapsed or refractory CLL/SLL or Non-Hodgkin's Lymphomas (escalation cohort), until the maximum tolerated dose or recommended dose is reached. Followed by up to 100 patients enrolled in the expansion cohort at the recommended dose.
  Interventions: Drug: CG-806

INTERVENTIONS:
Drug: CG-806 — CG-806 will be given orally in ascending doses starting at 150 mg PO BID until the maximum tolerated dose or recommended dose is reached.
  Other Names: Luxeptinib

SUMMARY:
This study is being done to evaluate the safety, tolerability and effectiveness of Oral CG-806 for the treatment of patients with chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), or Non-Hodgkin's Lymphomas who have failed or are intolerant to two or more lines of established therapy or for whom no other treatment options are available.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase Ia/b dose escalation study of safety, pharmacodynamics, and pharmacokinetics of CG-806 in ascending cohorts (3+3 design) to determine the MTD or recommended dose in patients with relapsed or refractory CLL/SLL or Non-Hodgkin's Lymphoma patients. This is to be followed by a cohort expansion phase at the MTD or recommended oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Life expectancy of at least 2 months
* ECOG Performance Status ≤ 2
* Patients must be able to swallow capsules
* Adequate hematologic parameters, unless cytopenias are disease caused
* Adequate renal, liver and cardiac function parameters

Exclusion Criteria:

* Patients with GVHD requiring systemic immunosuppressive therapy
* Uncontrolled leptomeningeal disease, auto-immune hemolytic anemia and uncontrolled and clinical significant disease related metabolic disorder
* Clinically significant intravascular coagulation
* Treatment with other investigational drugs within 14 days prior to first study treatment administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events of CG-806 | Cycle 1 (28 days)
  To determine the safety and tolerability of CG-806.
Establish a CG-806 dose that maintains a biologically active plasma concentration | Cycle 1 (28 days)
  To determine the dose of CG-806 given orally every 12 hours that maintains a biologically active plasma concentration over a period of 28 days.
Establish recommended dose for future development of CG-806 | Up to 10 months
  To establish the recommended Phase 2 dose (RP2D) of CG-806 for future clinical trials in patients with advanced CLL/SLL or NHL.

SECONDARY OUTCOMES:
Pharmacokinetic variables including maximum plasma concentration (Cmax) | Cycle 1 (28 days)
  Pharmacokinetic variables including maximum plasma concentration (Cmax)
Pharmacokinetic variables including minimum plasma concentration (Cmin) | Cycle 1 (28 days)
  Pharmacokinetic variables including minimum plasma concentration (Cmin)
Pharmacokinetic variables including Area Under the Curve (AUC) Pharmacokinetic variables including Area Under the Curve (AUC Pharmacokinetic variables including Area Under the Curve (AUC | Cycle 1 (28 days)
  Pharmacokinetic variables including Area Under the Curve (AUC)
Pharmacokinetic variables including volume of distribution | Cycle 1 (28 days)
  Pharmacokinetic variables including volume of distribution
Pharmacokinetic variables including clearance | Cycle 1 (28 days)
  Pharmacokinetic variables including clearance
Pharmacokinetic variables including serum half-life | Cycle 1 (28 days)
  Pharmacokinetic variables including serum half-life
To assess the antitumor activity of CG-806 using FDG PET-CT imaging evaluations | Average 2 Cycles (8 weeks)
  To assess the antitumor activity of CG-806 using FDG PET-CT imaging evaluations
Pharmacodynamic biomarkers of drug effect including BTK activity | Average 2 cycles (8 weeks)
  Pharmacodynamic biomarkers of drug effect including BTK activity
Pharmacodynamic biomarkers of drug effect including selected mRNA levels | Average 2 cycles (8 weeks)
  Pharmacodynamic biomarkers of drug effect including selected mRNA levels
To assess the relative BA of formulation G1 against formulation G2 | Cycle 1 (28 days)
  To assess the relative bioavailability of original formulation (G1) against new generation formulation (G2).
To assess the relative BA of formulation G1 against formulation G3 | Cycle 1 Lead-Up (3 days)
  To assess the relative bioavailability of original formulation (G1) against new generation formulation (G3).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Bejar, MD, PhD, Study Director — Aptose Biosciences Inc.
Locations (30):
- United States (30):
  - University of California Los Angeles, Los Angeles, California
  - Pacific Cancer Care, Monterey, California
  - Torrance Memorial Physician Network, Redondo Beach, California
  - UCSD Moores Cancer Center, San Diego, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - St. Joseph Heritage Heathcare, Santa Rosa, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - The Center for Cancer and Blood Disorders a division of American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - SCL Health, St. Vincent Frontier Cancer Center, Billings, Montana
  - Morristown Medical Center, Morristown, New Jersey
  - Manhattan Hematology Oncology, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Prisma Health - ITOR, Greenville, South Carolina
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - Texas Oncology - Austin-Midtown, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - University of Texas, M.D. Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, Mays Cancer Center, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, P.C. - Compass Oncology, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No